CLINICAL TRIAL: NCT03003936
Title: Glucose Tolerance, Meal Timing and MTNR1B in a Mediterranean Population
Brief Title: Glucose Tolerance, Meal Timing and MTNR1B
Acronym: ONTIME-DINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, PROF. MARTA GARAULET AZA, Full Proffesor, Universidad de Murcia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 15123/PI/10
Record Dates: First submitted 2016-12-16; First posted 2016-12-28 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Non-Diabetic Disorder of Endocrine Pancreas
Keywords: Glucose tolerance; MTNR1B; nutrigenomics; Food timing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Dinner Timing (Experimental): Test the lack of concurrence of meal timing with endogenous melatonin concentrations
  Interventions: Behavioral: Dinner timing
- Late Dinner Timing (Experimental): Test the concurrence of meal timing with elevated endogenous melatonin concentrations
  Interventions: Behavioral: Dinner timing

INTERVENTIONS:
Behavioral: Dinner timing — Glucose tolerance after a late diner (1 hour before habitual bedtime) differs from early dinner (4 hours before habitual bedtime) due to the concurrence of meal timing with different levels of endogenous melatonin. This effect can be different among risk allele carriers (G) or non-rick allele carriers (C) of the MTNR1B.

SUMMARY:
The purpose of this investigation is to assess in a community-based cohort of late-night eaters the effect of coincident food intake and endogenous melatonin on glycemic control, and the putative interaction effect of melatonin receptor 1B (MTNR1B) genetic variation on this relationship. With the results from this study, the investigators expect to advance in the understanding of the role of endogenous melatonin on glucose metabolism in late night eaters and carriers of the MTNR1B risk allele, with potential implications on the guidelines to mitigate risk of type 2 diabetes in late night eaters and carriers of the MTNR1B risk allele.

DETAILED DESCRIPTION:
Late-night dinner eating is associated with increased risk for type-2-diabetes. The underlying mechanism is unclear. One explanatory hypothesis is that the concurrence of elevated circulating melatonin and high glucose concentrations (characterizing late-eating) leads to impaired glucose-tolerance. However, to date, no study has tested the influence of physiological melatonin concentrations on glucose tolerance. The discovery of melatonin receptor MTNR1B as a diabetes risk gene provides evidence for a role of physiological levels of melatonin in glucose control.

The aim of the current study is to test the hypothesis that the concurrence of meal timing with elevated endogenous melatonin concentrations results in impaired glucose control and that this effect is stronger in homozygous MTNR1B risk carriers than in non-carriers. To do so we will test glucose tolerance using identical mixed meals under two dinner conditions: a) delayed dinner or Late Eating (LE): starting1 hour before usual bed time, b) advanced dinner or Early Eating (EE): starting 4 hours before habitual bed time, in a randomized, cross-over study design.

These findings could support a clinical application for the screening of this single nucleotide polymorphism (SNP) and the possibility of implementing tailored and cost-effective behavioral interventions to prevent type 2 diabetes in vulnerable populations.

These goals will be achieved through a specific approach:

• Interventional (randomized, cross-over controlled trials) (Aim 1): To study the potential interaction between meal timing (dinner) and genetic variants MTNR1B for glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: >19 kg/m2
* Age: >18 years of age
* Caucasian

Exclusion Criteria:

* Receiving treatment with thermogenic, lipogenic, or contraceptive drugs
* Diabetes mellitus, chronic renal failure, hepatic diseases, or cancer diagnosis
* Bulimia diagnosis, prone to binge eating
* Undergoing treatment with anxiolytic or antidepressant drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-12; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) glucose | between 0-120 minutes, Visit 2 and 3
  Investigators will measure glucose levels for 120 minutes at day time and night time visits, and compare the results by genotype at selected loci.

SECONDARY OUTCOMES:
Fasting glucose | between 0-120 minutes, Visit 2 and 3
Saliva Melatonin | between 0-120 minutes, Visit 2 and 3

OTHER OUTCOMES:
Sleep Duration | total of 2 weeks between Visit 1 and 3
  Sleep duration will be computed from self-reported.
Light Exposure | total of 2 weeks between Visit 1 and 3
  Measured using Pendant G Acceleration Data Logger.
Total Energy Intake | total of 2 weeks between Visit 1 and 3
  Total energy intake in kcal/day will be computed from 14-day 24-hr dietary record.
Dietary Composition | total of 2 weeks between Visit 1 and 3
  Macronutrient and micronutrient intake will be computed from 14-days of self-reported 24-hr dietary record.
Dietary Intake Timing | total of 2 weeks between Visit 1 and 3
  Food timing will be self-reported and averaged across 14-days of 24-hr dietary record.
Chronotype | at baseline
  Assessed using the Morningness-Eveningness Questionnaire (MEQ).

CONTACTS AND LOCATIONS:
Overall Officials: Marta Garaulet, PHD, Study Director — Universidad de Murcia
Locations (1):
- University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Minguez J, Saxena R, Bandin C, Scheer FA, Garaulet M. Late dinner impairs glucose tolerance in MTNR1B risk allele carriers: A randomized, cross-over study. Clin Nutr. 2018 Aug;37(4):1133-1140. doi: 10.1016/j.clnu.2017.04.003. Epub 2017 Apr 10. PMID 28455106